CLINICAL TRIAL: NCT05255679
Title: Pilot Study on the Effect of Early FES Cycling After Acute Spinal Cord Injury on Neuromuscular Preservation and Neurorecovery
Brief Title: Early FES Cycling in Acute Spinal Cord Injury for Neuromuscular Preservation and Neurorecovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Royal Alexandra Hospital (Other); Glenrose Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00100619
Record Dates: First submitted 2021-01-20; First posted 2022-02-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Spinal Cord Injury
Keywords: spinal cord injury; functional electrical stimulation; muscle mass; spasticity; neurorecovery
MeSH Terms: conditions — Spinal Cord Injuries; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: Non-randomized control group design
Who Masked: Outcomes Assessor
Masking Description: Person performing electrophysiology assessments will not know group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Early FES (Experimental): Receives standard care plus FES cycling in Phase 1 (starting 14 to 21 days after injury and for 3 months) and Phase 2 (from month 3 to month 6 after enrollment).
  Interventions: Device: Early FES
- Delayed FES (Experimental): Receives standard care only in Phase 1 (considered Control group in Phase 1), and standard care plus FES cycling in Phase 2 (from month 3 to month 6 after enrollment).
  Interventions: Device: Delayed FES
- Control (No Intervention): Receives standard care only

INTERVENTIONS:
Device: Early FES — FES cycling starting 14-21 days post SCI for 6 months, 3 sessions/week, with gradually increasing duration (15-60 minutes), cadence (20-45 RPM) and resistance; surface stimulation of 3-5 muscle groups per leg; with RT300 Supine or SLSA FES cycle (Restorative Therapies, Inc, Baltimore, MD)
  Arms: Early FES
Device: Delayed FES — FES cycling starting 3 months (+ 14-21 days) post SCI, for 3 months, 3 sessions/week, with gradually increasing duration (15-60 minutes), cadence (20-45 RPM) and resistance; surface stimulation of 3-5 muscle groups per leg; with RT300 Supine or SLSA FES cycle (Restorative Therapies, Inc, Baltimore, MD)
  Arms: Delayed FES

SUMMARY:
Spinal cord injury (SCI) is a devastating condition that often leads to paralysis and multiple health problems such as muscle wasting, bone loss and spasticity. Despite the paralysis, functional electrical stimulation (FES) on the skin surface muscles may produce muscle contractions. People who have had an SCI for a long time (chronic SCI) already use FES cycling to exercise, and it is known that it can reverse muscle atrophy and has a wide range of health benefits. Furthermore, animal research suggests that starting exercise training early after new SCI may promote spinal cord recovery. However, not much is known about early FES cycling in humans. Therefore, the investigators propose to study if early FES cycling could prevent muscle wasting, pain or spasticity, and help with spinal cord recovery.

The study will recruit 36 participants with a new, acute SCI, between 14 and 21 days after their injury into 3 groups. An Early-FES group starts FES cycling early after injury (between 14 and 21 days after injury), and for a duration of 6 months. A Delayed-FES group starts FES cycling 3 months after enrolling in the study, and for a duration of 3 months. A Control group does not perform FES cycling.

This pilot study will allow us to study if early FES cycling, in addition to normal care, has greater benefits on the preservation and recovery of the leg muscles and spinal cord function than delayed FES cycling or standard care only. The results of this pilot study may lead to the development of a larger study with early FES cycling after new SCI.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) usually results in weakness or paralysis in the legs and/or arms, depending on the level and severity of the damage to the spinal cord. In addition, people with SCI often develop several complications in the long term, such as muscle wasting (atrophy), loss of bone strength, pain, and spasticity.

Despite the weakness or paralysis, the muscles in a person with SCI can be activated using electrical stimulation applied on the skin surface of the muscles. This technique is called functional electrical stimulation (FES) and can be used in combination with a bike to perform a cycling movement (FES cycling). People who have had an SCI for a long time (chronic SCI) already use FES cycling to exercise, and it is known that it can reverse muscle atrophy and has a wide range of health benefits. Furthermore, animal research suggests that starting exercise training early after new SCI may promote spinal cord recovery. However, not much is known about early FES cycling in humans, for example, if it could prevent muscle atrophy, pain or spasticity, and help with recovery of the spinal cord. Therefore, the investigators propose to study if early FES cycling may prevent these complications and help with spinal cord recovery.

The study will recruit 36 participants with a new SCI, in 3 groups. The Early-FES group starts FES cycling early after injury (between 14 and 21 days after injury), and for a duration of 6 months. A Delayed-FES group starts FES cycling 3 months after enrolling in the study, and for a duration of 3 months. A Control group does not perform FES cycling. People with an acute, complete or incomplete SCI that resulted in paralysis from the waist down (paraplegia) or neck down (quadriplegia) will be considered. The Early and Delayed FES group will be recruited from the University of Alberta Hospital (UAH) where the FES bikes are available. Participants will be assigned by chance into Early and Delayed FES group. The control group will be mainly recruited from the Royal Alexandra Hospital, where the FES bikes are currently not available. The FES groups will perform FES cycling sessions 3 times per week (up to 1 hour per session) and receive standard care (typically including physical and occupational therapy). The Control group will only receive standard care.

The FES cycling will be performed while the participants are lying in bed using a bed bike, or while sitting in a wheel chair using chair-based bike. Both systems use pedals that are strapped to the feet and an electrical stimulator to activate several muscles of both legs using electrodes attached to the skin.

The following will be measured: 1) the size of the leg muscles and amount of fat in the legs using a CT scanner. 2) strength of the muscles using manual tests and by the electrical signals in the muscle. 3) spasticity by measuring electrical responses in the muscle when stimulated, as well as with clinical scales. 4) strength of the electrical connections between brain and spinal cord. 5) clinical measures such as the spinal injury classification, pain and reflexes. 6) response of participants to the FES cycling program. 7) cost and health care resources for the administration of early and delayed FES cycling. All 3 groups will undergo the same assessments.

This pilot study will allow the investigators to study if early FES cycling, in addition to standard care, has greater benefits on the preservation and recovery of the leg muscles and spinal cord function than standard care only. The results of this pilot study may lead to the development of a multi-center clinical trial with early FES cycling after new SCI, which may have important and innovative implications in the future rehabilitation practice, improving the health, function and quality of life of persons with SCI.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic or non-traumatic SCI
* Acute onset of SCI
* Able to start FES cycling 14-21 days post injury
* Injury level C1 - L5
* AIS A, B, C, D (ASIA Impairment Scale)
* Medically stable

Absolute Contraindications and Exclusion Criteria

1. AIS D, able to walk without assistive device
2. Unstable spine fractures
3. Unstable fractures/dislocations in lower extremities or pelvis
4. Pregnancy
5. Unable to give consent to participate in the study
6. Contraindications for TMS (Transcranial Magnetic Stimulation).

Relative Contraindications and Exclusion Criteria (Exclusion or Caution)

1. Lower motor neuron injury with insufficient muscle contraction with FES
2. Peripheral nerve or root injury resulting in denervated lower limb muscles
3. History of severe hip or knee instability or dislocation/subluxation
4. Osteoporosis in lower extremities that could result in fracture from cycling
5. Osteoarthritis in lower extremities
6. Limited range of motion in hip and knee preventing cycling
7. History of epilepsy not effectively managed by medication
8. History of heart problems (coronary artery disease / myocardial infarction / congestive heart failure)
9. Implanted cardiac demand pacemaker
10. Implanted stimulators: diaphragmatic, epidural, vagus nerve, phrenic
11. Malignant tumor in stimulated areas
12. Thrombophlebitis or thrombosis in stimulated area
13. Skin lesions or open wounds at any potential electrode site
14. Pressure ulcers that could deteriorate from cycling
15. Spasticity
16. Autonomic dysreflexia
17. Active heterotopic ossification in lower extremities
18. Extreme edema or adipose tissue in legs
19. Any other contraindications to participate in an active exercise program

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Muscle cross-sectional area thigh and calf: Change from 0 to 3 months | 3 months
  Muscle cross sectional area measured from multiple transverse CT scan slices across thigh and calf
Muscle cross-sectional area thigh and calf: Change from 3 months to 6 months | 3 months
  Muscle cross sectional area measured from multiple transverse CT scan slices across thigh and calf
Spasticity legs: Change from 0 to 3 months | 3 months
  Size of the cutaneomuscular reflex (CMR) produced by electrical stimulation of the medial arch of the foot and measured in the electromyogram (EMG) from several muscles in the leg (tibialis anterior, soleus, quadriceps and hamstrings).
Spasticity legs: Change from 3 months to 6 months | 3 months
  Size of the cutaneomuscular reflex (CMR) produced by electrical stimulation of the medial arch of the foot and measured in the electromyogram (EMG) from several muscles in the leg (tibialis anterior, soleus, quadriceps and hamstrings).
Corticospinal excitability: Change from 0 to 3 months | 3 months
  Size of the motor evoke potentials (MEP) produced by transcranial magnetic stimulation of the motor cortex, and measured in the EMG of several leg muscles (tibialis anterior, soleus, quadriceps and hamstrings).
Corticospinal excitability: Change from 3 months to 6 months | 3 months
  Size of the motor evoke potentials (MEP) produced by transcranial magnetic stimulation of the motor cortex, and measured in the EMG of several leg muscles (tibialis anterior, soleus, quadriceps and hamstrings).
Spinal cord excitability: Change from 0 to 3 months | 3 months
  Hmax/Mmax ratio, based on H-reflex and M-wave measurements in soleus EMG during tibial nerve stimulation, will be quantified as a measure of general spinal cord excitability (sensory transmission and motoneuron excitability)
Spinal cord excitability: Change from 3 months to 6 months | 3 months
  Hmax/Mmax ratio, based on H-reflex and M-wave measurements in soleus EMG during tibial nerve stimulation, will be quantified as a measure of general spinal cord excitability (sensory transmission and motoneuron excitability)
Muscle strength: Change from 0 to 3 months | 3 months
  Size of the EMG measured during maximum voluntary contraction in tibialis anterior, soleus, quadriceps and hamstrings.
Muscle strength: Change from 3 months to 6 months | 3 months
  Size of the EMG measured during maximum voluntary contraction in tibialis anterior, soleus, quadriceps and hamstrings.

SECONDARY OUTCOMES:
SCI Classification at Baseline | Baseline
  Spinal cord injury classification based on the American Spinal Injury Association (ASIA) Injury Scale (AIS), according to the International Standard for Neurological Classification of Spinal Cord Injury (ISNCSCI) exam. Range AIS A, B, C, D (most-least severe injury)
SCI Classification at 3 months | 3 months
  Spinal cord injury classification based on the American Spinal Injury Association (ASIA) Injury Scale (AIS), according to the International Standard for Neurological Classification of Spinal Cord Injury (ISNCSCI) exam. Range AIS A, B, C, D (most-least severe injury)
SCI Classification at 6 months | 6 months
  Spinal cord injury classification based on the American Spinal Injury Association (ASIA) Injury Scale (AIS), according to the International Standard for Neurological Classification of Spinal Cord Injury (ISNCSCI) exam. Range AIS A, B, C, D (most-least severe injury)
Motor scores: Change from 0 to 3 months | 3 months
  Sum of motor scores based on manual muscle strength testing of 5 key upper limb and 5 key lower limb muscle groups bilaterally according to the International Standard for Neurological Classification of Spinal Cord Injury (ISNCSCI) exam. Range worst-best score 0-100.
Motor scores: Change from 3 months to 6 months | 3 months
  Sum of motor scores based on manual muscle strength testing of 5 key upper limb and 5 key lower limb muscle groups bilaterally according to the International Standard for Neurological Classification of Spinal Cord Injury (ISNCSCI) exam. Range worst-best score 0-100.
Sensory scores: Change from 0 to 3 months | 3 months
  Sum of sensory scores in response to light touch and pinprick at 28 key sensory points on each side of the whole body, according to the International Standard for Neurological Classification of Spinal Cord Injury (ISNCSCI) exam. Range worst-best score 0-224.
Sensory scores: Change from 3 months to 6 months | 3 months
  Sum of sensory scores in response to light touch and pinprick at 28 key sensory points on each side of the whole body, according to the International Standard for Neurological Classification of Spinal Cord Injury (ISNCSCI) exam. Range worst-best score 0-224.
Pain intensity: Change from 0 to 3 months | 3 months
  Pain intensity assessment using the International Spinal Cord Injury Pain Basic Data Set v2. The tool scores intensity using an 11-point numeric scale (Range best-worst score 0-10). In addition the tool describes pain over the previous 7 days, impact of pain, type of pain (nociceptive vs. neuropathic), intensity and duration of pain, and treatment for pain.
Pain intensity: Change from 3 months to 6 months | 3 months
  Pain intensity assessment using the International Spinal Cord Injury Pain Basic Data Set v2. The tool scores intensity using an 11-point numeric scale (Range best-worst score 0-10). In addition the tool describes pain over the previous 7 days, impact of pain, type of pain (nociceptive vs. neuropathic), intensity and duration of pain, and treatment for pain.
Leg cross-sectional area thigh and calf: Change from 0 to 3 months | 3 months
  Leg cross-sectional area calculated based on circumferences of thigh and calf measured with tape measure, and corrected for skinfold thickness (measure of subcutaneous fat) measured with skinfold caliper at same locations.
Leg cross-sectional area thigh and calf: Change from 3 months to 6 months | 3 months
  Leg cross-sectional area calculated based on circumferences of thigh and calf measured with tape measure, and corrected for skinfold thickness (measure of subcutaneous fat) measured with skinfold caliper at same locations.
Walking Speed: Change from 0 to 3 months | 3 months
  Depending in the participant's capabilities, walking speed will be assessed with the 10-meter walking test (measuring time taken to walk 10 meters), and/or the 6-minute walking test (measuring distance walked in 6 minutes)
Walking Speed: Change from 3 months to 6 months | 3 months
  Depending in the participant's capabilities, walking speed will be assessed with the 10-meter walking test (measuring time taken to walk 10 meters), and/or the 6-minute walking test (measuring distance walked in 6 minutes)
Walking Capability: Change from 0 to 3 months | 3 months
  Scored using the Walking Index for Spinal Cord Injury (WISCI II), giving a ranking from most severe impairment (0) to least severe impairment (20) based on the use of devices, braces and physical assistance of one or more persons.
Walking Capability: Change from 3 months to 6 months | 3 months
  Scored using the Walking Index for Spinal Cord Injury (WISCI II), giving a ranking from most severe impairment (0) to least severe impairment (20) based on the use of devices, braces and physical assistance of one or more persons.
Spasticity self-report: Change from 0 to 3 months | 3 months
  Frequency and severity of the spasticity, its interference with function, and association with pain, scored using 11-point numeric scales. Range 0-10, with best (0) to worst (10).
Spasticity self-report: Change from 3 months to 6 months | 3 months
  Frequency and severity of the spasticity, its interference with function, and association with pain, scored using 11-point numeric scales. Range 0-10, with best (0) to worst score (10).
Depression at 3 months | 3 months
  Total score derived from the Patient Health Questionnaire (PHQ-9 ) which includes 9 questions related to signs of depression. Range best-worst score 0-27.
Depression at 6 months | 6 months
  Total score derived from the Patient Health Questionnaire (PHQ-9 ) which includes 9 questions related to signs of depression. Range best-worst score 0-27.
Psychosocial status of participants as assessed by AQol-8D at 3 months | 3 months
  Total score derived from the Assessment of Quality of Life (AQol-8D), measuring 8 dimensions of quality of life. Range worst-best score 35-176.
  Score derived from EQ-5D-5L Quality of Life Tool (EuroQol Research Foundation), measuring 5 dimensions. Range best-worst score 5-25.
Psychosocial status of participants as assessed by AQol-8D at 6 months | 6 months
  Total score derived from the Assessment of Quality of Life (AQol-8D), measuring 8 dimensions of quality of life. Range worst-best score 35-176.
  Score derived from EQ-5D-5L Quality of Life Tool (EuroQol Research Foundation), measuring 5 dimensions. Range best-worst score 5-25.
Program Cost | 6 months
  Cost and health care resources for the administration of early and delayed FES

CONTACTS AND LOCATIONS:
Overall Officials: Chester Ho, MD, Principal Investigator — University of Alberta; Monica A Gorassini, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No